CLINICAL TRIAL: NCT05771038
Title: Assessment of Bone Quality After Defective Socket Preservation Using Sodium Alendronate Gel Compared to Sticky Bone : A Histomorphometric Randomized Clinical Controlled Trial
Brief Title: Assessment of Bone Quality After Socket Preservation Using Sodium Alendronate Gel Compared to Sticky Bone
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Reda Hamed Elgohary, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sodiumalendronate ,stickybone
Record Dates: First submitted 2022-12-22; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Bone Quality Assessment; Preserved Sockets; Sodium Alendronate; Sticky Bone

STUDY DESIGN:
Intervention Model Description: * In first group: 20cc of venous blood is collected from the patient's forearm into silica-coated tube (10 ml) and 1 non coated vacutainer. Blood will be used to make injectable prf by spinning in centrifuge(2400-2700) for 2 minutes to produce autologous fibrin glue and then for 12 minutes+/- 2 minutes to obtain the concentrated growth factor layer. and sticky bone will be prepared then inserted into the socket.
  * In second group: prepared sodium alendronate gel will be placed in defective extraction sockets.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium alendronate group (Active Comparator): prepared sodium alendronate gel will be placed in defective extraction sockets.
  Interventions: Procedure: socket preservation using sodium alendronate gel
- stickybone group (Active Comparator): 20cc of venous blood is collected from the patient's forearm into silica-coated tube (10 ml) and 1 non coated vacutainer. Blood will be used to make injectable prf by spinning in centrifuge(2400-2700) for 2 minutes to produce autologous fibrin glue and then for 12 minutes+/- 2 minutes to obtain the concentrated growth factor layer. and sticky bone will be prepared then inserted into the socket.
  Interventions: Procedure: socket preservation using sticky bone

INTERVENTIONS:
Procedure: socket preservation using sodium alendronate gel — sockets will be preserved by sodium alendronate gel before then Patients will be evaluated after 3 days and weekly thereafter for the first month and then once monthly for signs of soft tissue irritation.
  After 3 months post-operative CBCT scans will be done to evaluate the bone density, alveolar crest bone height will be measured and core biopsy will be taken for Histomorphological study at the same visit where implant will be placed
  Arms: sodium alendronate group
Procedure: socket preservation using sticky bone — sockets will be preserved by sticky bone as mentioned before then Patients will be evaluated after 3 days and weekly thereafter for the first month and then once monthly for signs of soft tissue irritation.
  After 3 months post-operative CBCT scans will be done to evaluate the bone density, alveolar crest bone height will be measured and core biopsy will be taken for Histomorphological study at the same visit where implant will be placed
  Arms: stickybone group

SUMMARY:
The aim of study to evaluate the quality and quantity of the formed bone after socket preservation using sticky bone versus alendronate gel

DETAILED DESCRIPTION:
this study is alternative hypothesis research based on that one technique will be more efficient and effective than the other. In our case, the bone produced after introducing the sodium alendronate drug in defective sockets will be beneficial and will have better density and histomorphological features than treating the socket with sticky bone technique .

Several socket preservation techniques with different regenerative biomaterials and procedures as bone grafts, membranes, biological modifiers and platelet concentrates were introduced in the literature to overcome these problems.

Some researchers tried to introduce alternative techniques to preserve the socket depending on the enhancement of the native physiological mechanism of bone formation without the need for grafting through utilization of chemical agents that interfere with bone resorption, among these agents are the Bisphosphonates. Bisphosphonates are originally used in diseases with increased bone resorption as osteoporosis, paget's and fibrous dysplasia, hypercalcemia of malignancies.

The Effect of local delivery of alendronate on bone resorption following mucoperiosteal flap in mandible of rats was examined in Oxford Dental College Hospital, Bomannahalli on patients between 30 to 65 years old .and they found that alendronate reduces the resorptive activity of alveolar ridge significantly. It was found that local alendronate reduces active bone resorption without interfering with bone mineralization and quality. On remodeling surfaces local bisphosphonates binds to apatite crystals inhibiting their growth, aggregation and dissolution. As a result it decreases the turnover rate and increasing the mass and strength of bone.

Many authors as Jakobsen in 2009, supports the results from a study That found that the local Bisphosphonate (alendronate) treatment gives good bone quality and quantity.

So this study is conducted to evaluate the difference in bone quality and quantity produced on sockets preserved using sticky bone and local sodium alendronate compared to no intervention sockets.

Explanation for choice of comparators:

The main issue in traumatic Salama class 3 defective maxillary anterior sockets is the decreased amount of bone, sticky bone socket preservation technique needs venesection and it needs second surgical site adding more office time .on the other hand using sodium alendronate decreases the turnover rate and increasing the mass and strength of bone without the need of second surgical site or bone grafting material.

Clinical evaluation:

A through medical and dental history followed by clinical examination was carried out for all patients. Clinical measurements were taken to ensure patient adherence to our initial inclusion criteria prior to further investigations.

A pre-operative CBCT will be done to evaluate the height and the width of the intended alveolar ridge

Intra operative procedures for the study groups:

This clinical report describes Three different groups Following the protocol of The Oxford Dental College Hospital, Bomannahalli.

In all groups :

Infiltration anesthesia or nerve block according the socket were administered using mepivacaine HCl (2%) with levonordefrin 1:20 000 (Scandonest 2%; Septodont, Saint- Maur-des-Fossés, France). Injection to control pain and bleeding for hemostasis. Scrubbing and draping of the patient was carried out in a standard fashion using betadine , atraumatic extraction will then be done.

* In first group: 20cc of venous blood is collected from the patient's forearm into silica-coated tube (10 ml) and 1 non coated vacutainer. Blood will be used to make injectable prf by spinning in centrifuge(2400-2700) for 2 minutes to produce autologous fibrin glue and then for 12 minutes+/- 2 minutes to obtain the concentrated growth factor layer. and sticky bone will be prepared then inserted into the socket.
* In second group: prepared sodium alendronate gel will be placed in defective extraction sockets.

Follow up

Patients will be evaluated after 3 days and weekly thereafter for the first month and then once monthly for signs of soft tissue irritation.

After 3 months post-operative CBCT scans will be done to evaluate the bone density, alveolar crest bone height will be measured and core biopsy will be taken for Histomorphological study at the same visit where implant will be placed.

ELIGIBILITY:
Inclusion Criteria:

- defective class III sockets

* Patients with non-restorable teeth extracted sites
* Patients who have given their consent for this trial.
* Both genders males and females will be included.

Exclusion Criteria:

* Patients should not have taken drugs, especially bisphosphonates or drugs altering bone metabolism, within 2 months before the inclusion in the study.

  * Subjected to irradiation in the head and neck area less than 1 year before implantation.
  * Patients having history of allergy to any drugs.
  * Patients who have a history of any concomitant major known medical problem and/or ongoing pharmacologic treatments
  * Untreated periodontitis.
  * Poor oral hygiene and motivation.
  * Uncontrolled diabetes.
  * Pregnant or nursing.
  * Substance abuse.
  * Psychiatric problems or unrealistic expectations.
  * Severe bruxism or clenching.
  * Immunosuppressed or immunocompromised.
  * Treated or under treatment with intravenous amino-bisphosphonates.
  * Active infection or severe inflammation in the area intended for implant placement.
  * Unable to open mouth sufficiently to accommodate the surgical tooling.
  * Patients participating in other studies, if the present protocol could not be properly followed.
  * Referred only for implant placement or unable to attend a 5-year follow-up.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Histomorphometric analysis | 3 month from the socket preservation procedure
  bone sample will be taken and bone quality will be assesed

SECONDARY OUTCOMES:
Bone density | 3 month
  Bone density will be measured on CBCT
alveolar crest bone height | 3 month
  alveolar crest bone height will be measured on CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Saulacic N, Munoz F, Kobayashi E, Chappuis V, Gonzales-Cantalapiedra A, Hofstetter W. Effects of local application of alendronate on early healing of extraction socket in dogs. Clin Oral Investig. 2020 Apr;24(4):1579-1589. doi: 10.1007/s00784-019-03031-7. Epub 2019 Jul 26. PMID 31346723